CLINICAL TRIAL: NCT04691778
Title: Coronary Chronic Total Occlusion Percutaneous Coronary Intervention Using Antegrade Wiring Strategy With a First-choice Gladius Guidewire: a Randomized Clinical Study (Gladius First Trial)
Brief Title: Coronary CTO PCI Using Antegrade Wiring Strategy With a First-choice Gladius Guidewire (Gladius First)
Acronym: Gladius First
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2.59/III/20
Record Dates: First submitted 2020-12-18; First posted 2020-12-31 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-02

CONDITIONS: Coronary Artery Disease; Coronary Occlusion; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease; Coronary Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTO PCI using antegrade wiring strategy starting with the Gladius guidewire (Active Comparator): Study subjects will undergo CTO PCI with primary antegrade wiring strategy starting with the Gladius guidewire. In case of failed CTO crossing with the Gladius wire, the decision on continuing antegrade wire escalation with a different wire or switching to a different CTO PCI strategy will be left to the discretion of the operator.
  Interventions: Procedure: CTO PCI with the first-choice Gladius guidewire
- CTO PCI using standard antegrade wire escalation strategy (Other): Control subjects will undergo CTO PCI using standard antegrade wiring strategy starting with the lower/intermediate penetration force guidewires and, if necessary, escalating up to high gram-force guidewires, but without the use of first-choice Gladius guidewire.
  Interventions: Procedure: CTO PCI without the first-choice Gladius guidewire

INTERVENTIONS:
Procedure: CTO PCI with the first-choice Gladius guidewire — CTO PCI using antegrade wiring strategy with the first-choice Gladius guidewire
  Arms: CTO PCI using antegrade wiring strategy starting with the Gladius guidewire
Procedure: CTO PCI without the first-choice Gladius guidewire — CTO PCI using standard antegrade wire escalation strategy
  Arms: CTO PCI using standard antegrade wire escalation strategy

SUMMARY:
The Gladius First trial is designed as a single-centre, open, prospective, randomized clinical trial aimed to assess the efficiency and safety of coronary chronic total occlusion (CTO) percutaneous coronary intervention (PCI) using the antegrade wiring strategy with a first-choice intermediate Gladius guidewire. To this end, consecutive patients referred to CTO PCI with intended primary antegrade wire escalation strategy, will be randomized in a 1:1 fashion to antegrade wiring starting with the Gladius guidewire or antegrade wiring using the standard guidewire escalation strategy.

ELIGIBILITY:
Inclusion Criteria:

* delivery of an informed consent and compliance with study protocol
* CTO of a major coronary artery with at least intermediate difficulty score (J-CTO ≥1) as assessed by invasive angiography
* referral to clinically indicated CTO PCI with intended primary antegrade wiring strategy

Exclusion Criteria:

* in-stent CTO
* unstable angina and/or myocardial infarction
* prior myocardial infarction within 4 weeks before study enrolment
* CTO of a major coronary artery with an easy difficulty score (J-CTO 0) as assessed by invasive coronary angiography
* lack of valid antegrade wire escalation strategy as assessed by 2 independent CTO PCI operators
* chronic kidney disease (defined as eGFR ≤30 ml/min/m2)
* contraindication to antiplatelet therapy and/or heparin
* severe inflammatory disease
* positive pregnancy test or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
time-efficiency of antegrade wiring strategy | during procedure (intraprocedural)
  time-efficiency of antegrade wiring strategy defined as the time from advancement of the first wire into the proximal cap to either the time of successful antegrade wiring through the lesion or the time of cessation of antegrade wiring and changing CTO PCI strategy according to the hybrid algorithm

SECONDARY OUTCOMES:
time-efficiency of successful antegrade wiring strategy | during procedure (intraprocedural)
  time-efficiency of successful antegrade wiring strategy defined as the time from advancement of the first wire into the proximal cap to the time of successful antegrade wiring through the lesion
time-efficiency of successful antegrade approach | during procedure (intraprocedural)
  time-efficiency of successful antegrade approach defined as the time from advancement of the first wire into the proximal cap to either the time of successful antegrade wiring through the lesion or successful antegrade dissection and re-entry strategy
time-efficiency of antegrade approach | during procedure (intraprocedural)
  time-efficiency of antegrade approach defined as the time from advancement of the first wire into the proximal cap to either the time of successful antegrade wiring or antegrade dissection and re-entry strategy or the time of failed antegrade approach and changing CTO PCI strategy according to the hybrid algorithm
time-efficiency of successful CTO recanalization using any technique | during procedure (intraprocedural)
  time-efficiency defined as the time from advancement of the first wire into the proximal cap to the time of successful CTO recanalization using any technique (including antegrade and retrograde strategies)
total procedural time | during procedure (intraprocedural)
  total procedural time defined as the time from getting arterial access to the time of removal of the arterial sheaths
successful guidewire crossing through CTO using antegrade wiring strategy | during procedure (intraprocedural)
  successful guidewire crossing through CTO using antegrade wiring strategy
successful guidewire crossing through CTO with restoration of flow using antegrade wiring strategy | during procedure (intraprocedural)
  successful guidewire crossing through CTO with restoration of flow (<50% residual stenosis and TIMI flow grade 3) using antegrade wiring strategy
successful guidewire crossing through CTO using antegrade approach (including antegrade wiring and antegrade dissection and re-entry strategies) | during procedure (intraprocedural)
  successful guidewire crossing through CTO using antegrade approach (including antegrade wiring and antegrade dissection and re-entry strategies)
successful guidewire crossing through CTO with restoration of flow using antegrade approach (including antegrade wiring and antegrade dissection and re-entry strategies) | during procedure (intraprocedural)
  successful guidewire crossing through CTO with restoration of flow (<50% residual stenosis and TIMI flow grade 3) using antegrade approach (including antegrade wiring and antegrade dissection and re-entry strategies)
final procedural success defined as successful guidewire crossing through CTO with restoration of flow | during procedure (intraprocedural)
  final procedural success defined as successful guidewire crossing through CTO with restoration of flow (<50% residual stenosis and TIMI flow grade 3)
contrast volume related to successful guidewire crossing through CTO using antegrade wiring strategy | during procedure (intraprocedural)
  contrast volume related to successful guidewire crossing through CTO using antegrade wiring strategy
total contrast volume | during procedure (intraprocedural)
  total contrast volume
radiation dose related to successful guidewire crossing through CTO using antegrade wiring strategy | during procedure (intraprocedural)
  radiation dose related to successful guidewire crossing through CTO using antegrade wiring strategy
total radiation dose | during procedure (intraprocedural)
  total radiation dose
incidence of periprocedural complications | during hospitalization (assessed up to 30 days)
  incidence of periprocedural complications defined as: coronary perforation, tamponade, life-threatening arrhythmia requiring treatment, transient ischemic attack, stroke, myocardial infarction, urgent cardiac surgery, death

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Cardiology, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No